CLINICAL TRIAL: NCT01056185
Title: An International Observational Study to Characterize Adults Who Are Hospitalized With Influenza or Other Targeted Respiratory Viruses
Brief Title: Respiratory Virus Hospitalization Study (FLU 003 Plus)
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH); Clinical & Translational Science Institute, University of Minnesota (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0603M83587 FLU 003
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Influenza; Novel Respiratory Virus-1 Middle Eastern Respiratory Syndrome Coronavirus (MERS-CoV); Novel Respiratory Virus-2 Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)
Keywords: influenza; flu; swine flu; respiratory virus; hospitalization; MERS-CoV; SARS-CoV
MeSH Terms: conditions — Influenza, Human; Severe Acute Respiratory Syndrome; Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, respiratory for all participants. For participants with a confirmed targeted non-influenza respiratory virus, attempts will be made to obtain a sample of the local specimen used to confirm diagnosis.
  Whole blood for human genomics (only for FLU 003 Plus sites opting to also participate in INSIGHT Genomics and participant has signed an additional consent)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Influenza: Influenza A and subtypes such as H3N2 and 2009 H1N1 or influenza B
- Novel Respiratory Virus-1: MERS-CoV (Middle East Respiratory Syndrome Coronavirus
- Novel Respiratory Virus-2: SARS-CoV (Severe Acute Respiratory Syndrome Coronavirus)

SUMMARY:
Following the sudden and unexpected emergence of influenza A(H1N1)pdm09 (2009 H1N1) virus, this observational study was initiated to estimate rates of morbidity and mortality and to examine predictors of severity among participants with 2009 H1N1 infection. In 2011, as surveillance indicated that 2009 H1N1 virus was co-circulating with other seasonal influenza A and B viruses worldwide, the protocol was expanded to include other influenza A subtypes and influenza B viruses. The current version of the protocol (released in August 2013) further broadens the scope of this observational study. With the recognition that novel respiratory viruses other than novel influenza A viruses, e.g., Middle East Respiratory Syndrome Coronavirus (MERS-CoV), could become prevalent and of major public health importance, the objectives of this protocol have been expanded.

DETAILED DESCRIPTION:
The purpose of this observational study is to describe the characteristics and outcomes over a 60-day follow-up period of participants with influenza virus infection (including influenza A subtypes such as H3N2 and 2009 H1N1, or influenza B), or a targeted non-influenza respiratory virus, who are hospitalized with severe illness and/or complications in geographically diverse locations.

Specific objectives related to influenza virus infection are to estimate the percentage of participants who go on to develop severe disease or complications that require hospitalization; to obtain information on risk factors for disease severity; and to establish a central repository of specimens for use in virus characterization, including subtyping, antigenic and genetic analyses, identification of signature mutations associated with antiviral drug resistance, mutational evolution, and additional reassortment.

Specific objectives related to novel non-influenza respiratory viruses of potential major public health importance are to characterize initial cases and their outcomes in order to develop more specific protocols that could inform the prevention and treatment of these new infections.

The information used from this study on participants with influenza and novel respiratory virus infections will be rapidly analyzed and shared broadly in order to guide policymakers and to design future studies.

Approximately 500 patients with influenza will be enrolled each year at an estimated 75 sites which are in geographically diverse locations across several continents.

Study Plan:

* Participants who meet the eligibility criteria will be enrolled at participating clinical sites.
* Patients with a diagnosis of influenza (confirmed or suspected), who are hospitalized with complications or severe disease, will be enrolled.
* At enrollment, consent is signed and information (demographics, medical history (including prior influenza and pneumococcal vaccination), medications (including antivirals) and treatments prescribed) will be recorded. A blood sample for serum and plasma will be obtained at enrollment, as well as an upper respiratory tract sample and lower respiratory tract sample, if appropriate. The respiratory specimens will be sent for central reverse transcriptase polymerase chain reaction (RT-PCR) testing for influenza.
* For participants who are still hospitalized, and not intubated, 5 to 7 days after enrollment an additional upper respiratory sample is obtained.
* Status will be re-assessed at approximately 28 days and 60 days after enrollment and another blood sample for serum and plasma will obtained at both time points.
* For participants who are mechanically ventilated additional upper and lower respiratory tract specimens will be obtained at specific timepoints.

In February 2012, the FLU 004 Genomics protocol v 1.0 was released to the field. In August 2013, v 2.0 of the protocol was released as INSIGHT Genomics. The protocol was expanded beyond the FLU 002 and FLU 003 studies to include all qualifying INSIGHT studies (list of qualifying studies is posted on the INSIGHT website, www.insight-trials.org). The purpose of this substudy is to obtain a whole blood sample from which DNA will be extracted to study polymorphisms in immune response genes and other genetic variants that may be associated with an increased risk of severe influenza.

Participating FLU 003 Plus sites are given the option to also participate in INSIGHT Genomics which requires a separate protocol registration. Participants, once consented to FLU 003 Plus, will be offered the option to also consent to INSIGHT Genomics which includes a single whole blood sample collection. Participation in FLU 003 Plus will not be compromised if a participant opts not to participate in INSIGHT Genomics.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18 years of age
* Have been admitted to hospital
* Have a signed informed consent by participant or surrogate/representative
* Have a local diagnosis (confirmed or suspected) of influenza, or of a targeted non-influenza viral respiratory infection*, resulting in (or extending a previous) hospitalization

  * A list of targeted non-influenza respiratory viruses is maintained on the INSIGHT website.

Exclusion Criteria:

* Current imprisonment, or compulsory detention (involuntary incarceration) for treat of a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are hospitalized with a diagnosis (confirmed or suspected) of influenza or a targeted non-influenza viral respiratory infection, as soon as possible after the suspected diagnosis is made. Participants may have already been admitted to the hospital at the study site or may have been previously seen at another hospital where the diagnosis of influenza or infection with a targeted respiratory virus was made.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-08 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Death | 60-day period following enrollment

SECONDARY OUTCOMES:
Recovery from influenza illness (including days lost from normal activities) duration of hospitalization, days in intensive care, days of mechanical ventilation, days of dialysis, pregnancy outcome | approximately 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Cavan Reilly, PhD, Principal Investigator — University of Minnesota - Dept Biostatistics
Locations (63):
- United States (18):
  - UCSD Antiviral Research Center, San Diego, California
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - University of Illinois at Chicago, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cooper University Hospital, Camden, New Jersey
  - New Jersey Medical School Adult Clinical Research Center, Newark, New Jersey
  - Cornell ID-CRU, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - University of Tennessee College of Medicine, Chattanooga, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (11):
  - Hospital Nacional Profesor Alejandro Posadas, El Palomar, Buenos Aires
  - Instituto Medico Platense, La Plata, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Hospital Profesor Bernardo Houssay, Vicente López, Buenos Aires
  - Sanatorio Britanico, Rosario, Santa Fe Province
  - CEMIC, Buenos Aires
  - Hospital General de Agudos JM Ramos Mejia, Buenos Aires
  - Hospital Interzonal General de Agudos Dr. Diego Paroissien, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Hospital Rawson, Córdoba
- Australia (3):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- Centre Hospitalier Universitaire St. Pierre (C.H.U. St. Pierre), Brussels, Belgium
- Chile (2):
  - Clinica Alemana, Santiago
  - Fundacion Arriaran, Santiago
- Denmark (4):
  - Arhus Universitetshospital, Skejby, Aarhus
  - CHIP, Copenhagen
  - Hvidovre University Hospital, Department of Infectious Diseases, Hvidovre
  - Odense University Hospital, Odense
- Germany (3):
  - Medizinische Universitatsklinik - Bonn, Immunologische Ambulanz CRS, Bonn
  - Klinik I fur Innere Medizin der Universitat zu Koln, Studienburo fur Infektiologie u. HIV, Cologne
  - Johann Wolfgang Goethe - University Hospital, Infektionsambulanz CRS, Frankfurt
- Greece (4):
  - 1st Dept of Critical Care Medicine and Pulmonary Services, Evangelismos Hospital, Athens
  - 1st Respiratory Medicine Dept, Athens Hosp for Diseases of the Chest "Sotiria Hospital", Athens
  - Evangelismos General Hospital, Athens
  - Hippokration University General Hospital of Athens, Athens
- Peru (2):
  - Hospital Nacional Arzobispo Loayza, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
- Spain (5):
  - Hospital Clinico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Gregorio Mara�on, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Txagorritxu, Vitoria-Gasteiz
- Thailand (3):
  - Chulalongkorn University Hospital, Bangkok
  - Khon Kaen University, Srinagarind Hospital, Khon Kaen
  - Bamrasnaradura Institute, Nonthaburi
- United Kingdom (7):
  - Heatherwood and Wexham Park Hospitals NHS Foundation Trust, Slough, Berkshire
  - Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex
  - Churchill Hospital, Headington, Oxford
  - Sheffield Teaching Hospital NHS Foundation Trust, Sheffield, South Yorkshire
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, West Yorkshire
  - St James's University Hospital, Leeds, West Yorkshire
  - Newcastle General Hospital, Newcastle upon Tyne

REFERENCES:
- [Background] Novel Swine-Origin Influenza A (H1N1) Virus Investigation Team; Dawood FS, Jain S, Finelli L, Shaw MW, Lindstrom S, Garten RJ, Gubareva LV, Xu X, Bridges CB, Uyeki TM. Emergence of a novel swine-origin influenza A (H1N1) virus in humans. N Engl J Med. 2009 Jun 18;360(25):2605-15. doi: 10.1056/NEJMoa0903810. Epub 2009 May 7. PMID 19423869
- [Background] World Health Organization (WHO), www.who.int/, accessed 26 August 2013
- [Background] Guery B, Poissy J, el Mansouf L, Sejourne C, Ettahar N, Lemaire X, Vuotto F, Goffard A, Behillil S, Enouf V, Caro V, Mailles A, Che D, Manuguerra JC, Mathieu D, Fontanet A, van der Werf S; MERS-CoV study group. Clinical features and viral diagnosis of two cases of infection with Middle East Respiratory Syndrome coronavirus: a report of nosocomial transmission. Lancet. 2013 Jun 29;381(9885):2265-72. doi: 10.1016/S0140-6736(13)60982-4. Epub 2013 May 30. PMID 23727167
- [Background] Drosten C, Seilmaier M, Corman VM, Hartmann W, Scheible G, Sack S, Guggemos W, Kallies R, Muth D, Junglen S, Muller MA, Haas W, Guberina H, Rohnisch T, Schmid-Wendtner M, Aldabbagh S, Dittmer U, Gold H, Graf P, Bonin F, Rambaut A, Wendtner CM. Clinical features and virological analysis of a case of Middle East respiratory syndrome coronavirus infection. Lancet Infect Dis. 2013 Sep;13(9):745-51. doi: 10.1016/S1473-3099(13)70154-3. Epub 2013 Jun 17. PMID 23782859
- [Background] World Health Organization (WHO), Severe Acute Respiratory Syndrome (SARS), www.who.int/csr/sars/, accessed 26 August 2013
- [Derived] Wendt CH, Castro-Pearson S, Proper J, Pett S, Griffin TJ, Kan V, Carbone J, Koulouris N, Reilly C, Neaton JD; INSIGHT FLU003 Plus Study Group. Metabolite profiles associated with disease progression in influenza infection. PLoS One. 2021 Apr 2;16(4):e0247493. doi: 10.1371/journal.pone.0247493. eCollection 2021. PMID 33798209
- [Derived] Simonsen L, Higgs E, Taylor RJ, Wentworth D, Cozzi-Lepri A, Pett S, Dwyer DE, Davey R, Lynfield R, Losso M, Morales K, Glesby MJ, Weckx J, Carey D, Lane C, Lundgren J; INSIGHT FLU002 and FLU003 Study Groups. Using Clinical Research Networks to Assess Severity of an Emerging Influenza Pandemic. Clin Infect Dis. 2018 Jul 18;67(3):341-349. doi: 10.1093/cid/ciy088. PMID 29746631
- [Derived] Pett SL, Kunisaki KM, Wentworth D, Griffin TJ, Kalomenidis I, Nahra R, Montejano Sanchez R, Hodgson SW, Ruxrungtham K, Dwyer D, Davey RT, Wendt CH; INSIGHT FLU003 Plus Study Group. Increased Indoleamine-2,3-Dioxygenase Activity Is Associated With Poor Clinical Outcome in Adults Hospitalized With Influenza in the INSIGHT FLU003Plus Study. Open Forum Infect Dis. 2017 Oct 25;5(1):ofx228. doi: 10.1093/ofid/ofx228. eCollection 2018 Jan. PMID 29322062
- [Derived] Lynfield R, Davey R, Dwyer DE, Losso MH, Wentworth D, Cozzi-Lepri A, Herman-Lamin K, Cholewinska G, David D, Kuetter S, Ternesgen Z, Uyeki TM, Lane HC, Lundgren J, Neaton JD; INSIGHT Influenza Study Group. Outcomes of influenza A(H1N1)pdm09 virus infection: results from two international cohort studies. PLoS One. 2014 Jul 8;9(7):e101785. doi: 10.1371/journal.pone.0101785. eCollection 2014. PMID 25004134
- See also: INSIGHT website — http://www.insight-trials.org